CLINICAL TRIAL: NCT07331246
Title: Transcutaneous Electrical Nerve Stimulation (TENS) for Pain Relief During Transperineal MRI-Ultrasound Fusion-Guided Prostate Biopsy: An Exploratory Single-Center, Randomized, Placebo-Controlled Trial
Brief Title: TENS for Pain Relief During Fusion-Guided Prostate Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Bartłomiej Marczak, MD, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KB/531/2023, KB/531-116/2025
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Prostate Biopsy; Fusion Biopsy; Pain Management
MeSH Terms: conditions — Prostatic Neoplasms; Agnosia | interventions — Transcutaneous Electric Nerve Stimulation; Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A. Local Anesthesia Only (Control Group) (Active Comparator): Participants receive standard local anesthesia for transperineal MRI-ultrasound fusion-guided prostate biopsy using 1% lignocaine (20 mL total). No additional intervention is applied.
  Interventions: Procedure: Local Anesthesia
- B. TENS + Local Anesthesia (Experimental): Participants receive transcutaneous electrical nerve stimulation (TENS) applied to the perineum in addition to standard local anesthesia.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS); Procedure: Local Anesthesia
- C. Sham TENS + Local Anesthesia (Placebo Comparator): Participants receive sham (inactive) TENS with standard local anesthesia. Electrodes are applied as in Group B, but no electrical stimulation is delivered.
  Interventions: Device: Sham Transcutaneous Electrical Nerve Stimulation (Sham TENS); Procedure: Local Anesthesia

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Application of transcutaneous electrical nerve stimulation (TENS) using two pairs of adhesive electrodes placed in the perineal region. Electrical stimulation was initiated 3-5 minutes before local anesthetic infiltration and continued throughout the biopsy procedure. The device used symmetrical biphasic pulses at 80 Hz with a pulse width of 180 μs. Amplitude was adjusted to the maximum comfortable level for each participant. All participants underwent transperineal MRI-ultrasound fusion-guided prostate biopsy under local anesthesia. The study evaluated the effect of active versus sham transcutaneous electrical nerve stimulation (TENS) as an adjunct to pain management during the procedure.
  Other Names: TENS Therapy; Electrical Nerve Stimulation
  Arms: B. TENS + Local Anesthesia
Device: Sham Transcutaneous Electrical Nerve Stimulation (Sham TENS) — Application of sham transcutaneous electrical nerve stimulation (TENS) using identical electrode placement and device setup as the active TENS group, but without delivery of electrical current. The device was powered on but modified to prevent active stimulation. Participants were not informed of the inactive nature of the intervention. All participants underwent transperineal MRI-ultrasound fusion-guided prostate biopsy under local anesthesia. The study evaluated the effect of active versus sham transcutaneous electrical nerve stimulation (TENS) as an adjunct to pain management during the procedure.
  Other Names: Sham TENS; Placebo TENS; Inactive Electrical Stimulation
  Arms: C. Sham TENS + Local Anesthesia
Procedure: Local Anesthesia — Administration of 1% lignocaine (20 mL total) using a full needle path technique for anesthesia of the perineal skin and periprostatic tissue. No TENS electrodes or placebo stimulation applied. This represents standard of care anesthesia during transperineal MRI-ultrasound fusion-guided prostate biopsy.
  Other Names: Perineal Infiltration and Periprostatic Nerve Block; Standard Transperineal Local Anesthesia

SUMMARY:
The goal of this clinical trial is to learn whether transcutaneous electrical nerve stimulation (TENS) can reduce pain during transperineal prostate biopsy in adult male patients. It will also assess the safety and tolerability of using TENS in this setting. The main questions it aims to answer are:

Does TENS lower patient-reported pain during local anesthesia and prostate biopsy sampling?

Are there any side effects or complications associated with using TENS during the procedure?

Researchers will compare TENS to a placebo (sham TENS with no active stimulation) and to standard care (local anesthesia alone).

Participants will:

Be randomly assigned to receive either TENS + local anesthesia, sham TENS + local anesthesia, or local anesthesia alone

Undergo a standard transperineal prostate biopsy guided by MRI-ultrasound fusion

Report their pain levels during four specific stages of the procedure

Attend a follow-up visit 3-4 weeks after the biopsy to review results and assess for any side effects

ELIGIBILITY:
Inclusion Criteria:

* Suspicious lesions on multiparametric MRI, classified as PI-RADS score ≥ 3
* The indication for mpMRI was based on the presence of at least one of the following:
* Elevated serum prostate-specific antigen (PSA) levels
* Abnormal digital rectal examination (DRE)

Exclusion Criteria:

* Prior treatment of prostate cancer
* Contraindications to TENS, including:

  * Cutaneous damage or dermatologic conditions at the TENS application sites
  * Presence of cardiac pacemakers or automatic implantable cardioverter-defibrillators (AICDs)
  * Uncontrolled cardiac arrhythmias or congestive heart failure
  * History of epilepsy or seizure disorders
  * Metal implants near the site of stimulation
  * Malignancy at or near the site of stimulation
* Contraindications to transperineal biopsy, including:

  * Active urinary tract infection
  * Bleeding disorders or ongoing anticoagulant therapy
  * Anatomical abnormalities that prevent safe access to the prostate
* Known allergy or intolerance to local anesthetics or biopsy-related materials
* Severe comorbidities or unstable medical conditions that could compromise procedural safety
* Inability to provide informed consent or refusal to sign the consent form

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male participants only. Eligibility is limited to individuals assigned male at birth due to the requirement for a prostate.
Enrollment: 84 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity during transperineal prostate biopsy | Immediately after each procedural stage (within 30 seconds)
  Pain will be measured using the Numeric Rating Scale (0 = no pain, 10 = worst imaginable pain) at four key stages of the procedure: (1) ultrasound probe insertion, (2) perineal skin infiltration, (3) peri-prostatic nerve block, and (4) biopsy sampling.

SECONDARY OUTCOMES:
Incidence of adverse events related to biopsy or TENS application | Up to 30 days after biopsy
  All adverse events will be recorded, including skin irritation, discomfort, bleeding, urinary retention, or infection. Events will be classified using the Clavien-Dindo system.
Participant perception of TENS activity (blinding assessment) | Immediately after the procedure
  After the procedure, participants in the TENS or sham groups will be asked whether they believed the TENS device was active. Responses will be used to evaluate the effectiveness of participant blinding.
Correlation between number of biopsy cores and pain score | Immediately after biopsy sampling
  Spearman correlation will be used to assess whether the number of biopsy cores taken per lesion is associated with increased patient-reported pain during the sampling phase of the biopsy procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Medical University of Gdansk, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) to be shared will include:
  De-identified participant-level data relevant to primary and secondary outcome measures
  Pain score responses at each procedural stage (Numeric Rating Scale data)
  Group assignment (active TENS, sham TENS, or control)
  Adverse event data (Clavien-Dindo classification)
  Demographic and baseline clinical data (age, PSA level, BMI, prostate volume)
  No identifying information (e.g., names, birth dates, or hospital IDs) will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD and related documents will be available immediately after publication and will remain available for 5 years.
Access Criteria: Access will be granted to researchers with methodologically sound proposals for use in meta-analyses or individual participant data analyses. Data will be shared via a secure institutional repository after review and approval by the corresponding author.
URL: https://osf.io/jmuth